CLINICAL TRIAL: NCT01733589
Title: Multicenter Phase I/II Clinical Trial of Recombinant Human Endostatin Continued Pumping Into Vein Combining With Concurrent Chemo-Radiotherapy in the Patients With Unresectable Stage III Non-small-Cell Lung Cancer
Brief Title: Recombinant Human Endostatin Continued Pumping Into Vein Combining With CCRT in Unresectable Stage III NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Fudan University (Other); Peking University Cancer Hospital & Institute (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Shandong Cancer Hospital and Institute (Other); Jiangsu Cancer Institute & Hospital (Other); Fujian Cancer Hospital (Other Government); The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2012]-10-24
Record Dates: First submitted 2012-11-02; First posted 2012-11-27 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Stage III Non-small-Cell Lung Cancer
Keywords: Recombinant human endostatin; Non-small-Cell Lung Cancer; chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant Human Endostatin (Experimental): All patients received recombinant human endostatin(7.5mg/m2/24h) Continued Pumping Into Vein through 5 days at week 1, 3, 5, and 7. During week 2 through 8, patients received etoposide 50mg/m2 days 1-5 and cisplatin 50mg/m2 on day 1,8, every 4 weeks for two cycles with concurrent thoracic radiation at 60~66Gy in 30~33 fractions for 6~7 weeks.
  Interventions: Drug: Recombinant human endostatin; Drug: Etoposide (50mg/m2) IV (in the vein) on day 1 to day 5 of a 28-day cycle for 2 cycles; Drug: cisplatinum (50mg/m2) IV (in the vein) on day 1 and day 8 of a 28-day cycle for 2 cycles; Other: laboratory biomarker analysis; Other: CT perfusion imaging

INTERVENTIONS:
Drug: Recombinant human endostatin — Recombinant human endostatin(7.5mg/m2/24h) Continued Pumping Into Vein through 5 days at week 1, 3, 5, and 7,combined with concurrent chemo-radiotherapy.
Drug: Etoposide (50mg/m2) IV (in the vein) on day 1 to day 5 of a 28-day cycle for 2 cycles
Drug: cisplatinum (50mg/m2) IV (in the vein) on day 1 and day 8 of a 28-day cycle for 2 cycles
Other: laboratory biomarker analysis
Other: CT perfusion imaging

SUMMARY:
Resistance of hypoxic tumor cells to radiation is a significant reason of failure in the local control of tumors, especially the squamous cell carcinomas. Preclinical models have shown that Endostar may transiently "normalize" the tumor vasculature to make it more efficient for oxygen delivery, thereby providing a window of opportunity for enhanced sensitivity to radiation treatment. This study is to evaluate the safety, toxicity, and efficacy of the addition of Endostar Continued Pumping into Vein to the standard CCRT regimen in patients with unresectable stage III NSCLC.

DETAILED DESCRIPTION:
Primary

Evaluate the efficacy and safety of Endostar combined with concurrent chemo-radiotherapy (CCRT) in patients with unresectable stage III non-small-cell lung cancer (NSCLC).

Secondary

Measure changes in VEGF and other angiogenic cytokines and antiangiogenic factors in plasma samples from these patients.

Evaluate the application of CT perfusion imaging to determine changes in tumor vascular mophology and function during treatment.

ELIGIBILITY:
Inclusion Criteria:

* untreated histologic or cytologic of NSCLC verified
* inoperable stage IIIA or IIIB NSCLC
* measurable disease by RECIST
* 18~70 years of age
* an ECOG PS of 0 to 1
* absolute neutrophil count (ANC) of ≥1500/μL, hemoglobin ≥10gm/dL, platelet ≥100,000/μL
* serum creatinine ≤1.25 times of upper limit of normal (ULN), calculated creatinine clearance (CrCl) of ≥60ml/min
* bilirubin 1.5×ULN, AST and ALT less than 2.5×ULN, alkaline phosphatase less than 5×ULN
* forced vital capacity in 1 second (FEV1) higher than 0.8 L
* CB6 is normal
* Written informed consent

Exclusion Criteria:

* a history of other malignant diseases
* any contraindications for chemoradiotherapy
* distant metastasis
* malignant pleural and/or pericardial effusion
* pregnant or nursing
* preexisting bleeding diatheses or coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 2-year
  from beginning treatment to progressive disease or the last follow-up

SECONDARY OUTCOMES:
Response rate | 1 month
  complete response(CR); partial response(PR); stable disease(SD); progressive disease(PD)
overall survival | 5 years
  from date of beginning treatment until date of death
treatment related toxicities | 3 months
  radiation-induced esophagitis; radiation-induced pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China